CLINICAL TRIAL: NCT06579430
Title: Diagnostic Accuracy Study of Indocyanine Green for Perfusion Assessment
Acronym: Pre-CLOVER
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Erasmus Medical Center (Other); Leiden University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 201900307
Record Dates: First submitted 2024-08-21; First posted 2024-08-30 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Hypoparathyroidism
MeSH Terms: conditions — Hypoparathyroidism | interventions — Root Cause Analysis

STUDY DESIGN:
Intervention Model Description: A multicenter study is being conducted using standardized ICG-NIRF imaging of the parathyroid glands following total thyroidectomy. Perfusion curves are generated and analyzed postoperatively, with flow parameters being linked to postoperative parathyroid function.
  The study consists of two groups: the first group includes patients undergoing total thyroidectomy, where perfusion curves are compared between different patients. The second, smaller group is part of a root cause analysis, where the effects of injection speed and ICG concentration on the reproducibility of perfusion curves are evaluated by comparing curves within the same patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multicenter cohort (Experimental): Patients undergoing total thyroidectomy are included in this arm. Patients are included in the University Medical Center Groningen and the Erasmus Medical Center Rotterdam. After total thyroidectomy, the perfusion in the parathyroid glands is imaged utilizing ICG-NIRF. Postoperatively; perfusion curves are drawn for each parathyroid gland. Perfusion parameters are compared between patients and correlated to postoperative parathyroid function (PTH).
  Interventions: Drug: Indocyanine Green near infrared fluorescence imaging
- Root cause analysis (Experimental): Patients undergoing total or hemi-thyroidectomy are included in this arm. Patients are included in the University Medical Center Groningen. After (total/hemi)thyroidectomy, the perfusion in the parathyroid glands is imaged utilizing ICG-NIRF. A second measurement is performed in order to compare the influence of injection speed, camera and ICG dose on the curves. Postoperatively; perfusion curves are drawn for each parathyroid gland. Perfusion parameters are compared between the two measurements in the same patient.
  Interventions: Drug: Indocyanine Green near infrared fluorescence imaging

INTERVENTIONS:
Drug: Indocyanine Green near infrared fluorescence imaging — ICG-NIRF was performed using the Quest Spectrum Platform 2.0. The camera lens was positioned at a fixed distance of 30 cm to the wound bed, at a perpendicular angle, with the gain set at 22.5 decibels (dB) and an exposure time of 50 milliseconds (ms). ICG was dissolved in sterile water at a concentration of 2.5 mg/mL as recommended by the manufacturer (Verdye). 1.5 mg of ICG per liter of circulating blood volume was then administered through manual bolus intravenous injection. Blood volume estimation was based on the patient's height and weight.
  Other Names: Multicenter cohort
  Arms: Multicenter cohort
Drug: Indocyanine Green near infrared fluorescence imaging — ICG-NIRF was performed using the Quest Spectrum Platform 2.0. The camera lens was positioned at a fixed distance of 30 cm to the wound bed, at a perpendicular angle, with the gain set at 22.5 decibels (dB) and an exposure time of 50 milliseconds (ms). ICG was dissolved in sterile water at a concentration of 0.5 or 2.5 mg/mL as recommended by the manufacturer. 1.5 mg of ICG per liter of circulating blood volume was then administered through manual bolus intravenous injection. Blood volume estimation was based on the patients height and weight. Different administration rates (fast: 2s, slow: 15-20s) and a different camera system were tested.
  Group 1: Quest Platform 2.0; Fast/Slow; 2.5 mg/mL Group 2: Quest Platform 2.0; Slow/Fast; 2.5 mg/mL Group 3: Quest Platform 2.0; Fast/Fast; 2.5 mg/mL Group 4: Stryker Spy-Elite; Fast/Fast; 2.5 mg/mL Group 5: Quest Platform 2.0; Fast/Fast; 0.5 mg/mL
  Other Names: Root cause analysis
  Arms: Root cause analysis

SUMMARY:
Background Near-infrared fluorescence guided surgery with indocyanine green (ICG) was introduced for parathyroid perfusion assessment during total thyroidectomy in 2016. ICG can visualize tissue perfusion, since it becomes completely and permanently fixed to plasma proteins in the bloodstream, and circulates in the intravascular compartment only. ICG was already approved in 1956 for clinical use of tissue perfusion. However, until now there is still no (parathyroid) universal standard imaging protocol for ICG-guided fluorescent surgery including quantitative evaluation.

Main research question To develop a standardized universal imaging protocol for the assessment of parathyroid perfusion during total thyroidectomy with ICG including quantitative evaluation of the fluorescent signal.

• Design (including population, confounders/outcomes) This will be a proof-of-concept, prospective cohort study of patients undergoing an ICG-guided fluorescent total thyroidectomy to evaluate parathyroid gland perfusion. The main study endpoint is quantification of the fluorescent signal of ICG stratified by the occurrence of hypoparathyroidism. Hypoparathyroidism will be defined as a decrease in PTH of >70% at the first postoperative day. Furthermore, we will calculate the sensitivity of our model for the prediction of hypoparathyroidism.

Secondary outcomes are data from surgery, pre- and postoperative lab values (including calcium, PTH, albumin) and postoperative medication use.

Expected results We expect that the results of this study will lead to the development of a universal standard imaging protocol for ICG-guided fluorescent total thyroidectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Patients undergoing ICG-guided total thyroidectomy as surgical procedure for thyroid cancer, Graves' disease or goiter
3. Patients are eligible for surgery
4. Patients are mentally competent
5. Written informed consent

Exclusion Criteria:

1. Patients with known allergy for ICG or iodinated contrast
2. Pregnant or lactating women
3. Patients with previous neck surgery
4. Patients with dialysis dependent renal failure and kidney transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
Injection speed | During surgery
  The impact of injection speed on a parathyroid perfusion curve (slow vs fast)
ICG concentration | During surgery
  The impact of ICG concentration on a parathyroid perfusion curve (2.5 mg/mL vs 0.5 mg/mL)
Camera system | During surgery
  The impact of a camera system on a parathyroid perfusion curve (Quest vs SpyElite)

SECONDARY OUTCOMES:
Multicenter application | From surgery until one day post-surgery
  The correlation between postoperative hypoparathyroidism and the perfusion curve in two different centers (UMCG/EMC)

CONTACTS AND LOCATIONS:
Overall Officials: Schelto Kruijff, Professor, Principal Investigator — University Medical Center Groningen
Locations (2):
- Netherlands (2):
  - University Medical Center Groningen, Groningen
  - Erasmus Medical Center Rotterdam, Rotterdam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Noltes ME, Metman MJH, Jansen L, Peeperkorn EWM, Engelsman AF, Kruijff S. Parathyroid Function Saving Total Thyroidectomy Using Autofluorescence and Quantified Indocyanine Green Angiography. VideoEndocrinology. 2021 Jun 10;8(2):ve.2021.0008. doi: 10.1089/ve.2021.0008. eCollection 2021. PMID 34179223
- [Background] Noltes ME, Metman MJH, Heeman W, Rotstein L, van Ginhoven TM, Vriens MR, Engelsman AF, Boerma EC, Brouwers AH, van Dam GM, Pasternak JD, Kruijff S. A Novel and Generic Workflow of Indocyanine Green Perfusion Assessment Integrating Standardization and Quantification Toward Clinical Implementation. Ann Surg. 2021 Dec 1;274(6):e659-e663. doi: 10.1097/SLA.0000000000004978. PMID 34145192
- See also: Related Info — https://www.omig.nl/pre-clover/